CLINICAL TRIAL: NCT05351853
Title: Metabolic Effects of Plant-based Diet on Healthy Young Adults
Brief Title: Metabolic Effects of Plant-based Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 28041993
Record Dates: First submitted 2021-12-08; First posted 2022-04-28 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Healthy Diet; Fatty Liver; Insulin Resistance; Metabolic Syndrome; Healthy Lifestyle; Healthy Nutrition
Keywords: plant-based; metabolic; fatty-liver
MeSH Terms: conditions — Fatty Liver; Insulin Resistance; Metabolic Syndrome | interventions — Control Groups; Diet, Vegetarian; Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): 20 healthy individual will be in the control group. Participants of control group will not change their diet and will continue omnivore diet.
  Interventions: Dietary Supplement: Omnivore
- Vegetarian (Other): 20 healthy individual will be in the control group. Participants of this group will change their diet from omnivore to vegetarian (no meat /meat products) after the beginning of the study.
  Interventions: Dietary Supplement: Vegetarian
- Vegan (Other): 20 healthy individual will be in the control group. Participants of this group will change their diet from omnivore to vegan (%100 plant based) after the beginning of the study.
  Interventions: Dietary Supplement: Vegan

INTERVENTIONS:
Dietary Supplement: Omnivore — This study will evaluate effects of plant based diets (vegan and vegetarian). 60 omnivore individuals will be included. 20 of the participants will continue their omnivore diet as control group. 20 of the participants will change their diet to vegetarian, and 20 of them will change their diet to vegan.
  Other Names: Control Group
  Arms: Control Group
Dietary Supplement: Vegetarian — 20 of the participants will change their diet to vegetarian diet. In this group participants will not eat any meat or meat product but can eat/drink milk products, egg and other animal products.
  Arms: Vegetarian
Dietary Supplement: Vegan — 20 of the participants will change their diet to vegan diet. In this group participants will not eat any kind of animal products.
  Arms: Vegan

SUMMARY:
The purpose of this study is to assess the metabolic effects of plant based diet on healthy young adults.

DETAILED DESCRIPTION:
An internet announcement will be made and 60 participants who meet the eligibility requirements will be randomly selected. After being informed about study, all participants (60 omnivores) giving written informed consent will be assigned to the vegan and vegetarian groups of the study according to their preferences, while 20 participants will continue to be omnivores as the control group. At week 0 and 24, blood samples, urine samples, proton density fat fraction MRI evaluations and body composition analyze will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18-40 years old,
2. BMI is 18-30 kg/m2,
3. Having no chronic diseases,
4. Not smoking

Exclusion Criteria:

1. Having chronic disease,
2. Being older than 40 years old or younger than 18 years old,
3. Smoking,
4. Alcoholism or drinking more than 140 gr/week of alcohol,

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Liver Steatosis at 6 months | At week 24 liver steatosis change will be compared between the groups.
  Liver steatosis change will be compared between groups at the end of the study.

SECONDARY OUTCOMES:
Change from Baseline Insulin Resistance at 6 months | At week 24 insulin resistance change will be compared between the groups.
  Insulin resistance change will be compared between groups at the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University Medical Faculty, Istanbul, Turkey (Türkiye)